CLINICAL TRIAL: NCT06124508
Title: GUIAR: PromotinG Lung Cancer screenIng Awareness and Implementation in Hispanics/Latinx Head and Neck canceR Survivors
Brief Title: PromotinG Lung Cancer screenIng Awareness and Implementation in Hispanics/Latinx Head and Neck canceR Survivors
Acronym: GUIAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: LUNGevity Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Coral Olazagasti, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 20220746; K12CA226330 (NIH)
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: All participants will be randomized in a 1:1 ratio to the intervention or control arm via a blinded systematic randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Cancer Screening Education Group (Experimental): Participants in this group will receive intensive lung cancer screening and tobacco cessation education for up to two years.
  Interventions: Behavioral: Lung Cancer Screening Education; Behavioral: Semi-Structured Interview; Behavioral: Standard of Care Lung Cancer Screening Program
- Standard of Care Control Group (Other): Participants in this group will receive the standard of care treatment for up to two years.
  Interventions: Behavioral: Standard of Care Lung Cancer Screening Program

INTERVENTIONS:
Behavioral: Lung Cancer Screening Education — Tailored lung cancer screening education will consist of an annual, in-person 60 minute visit of lung cancer screening education in the participant's native language with material in layman's terms about the importance of lung cancer screening, tobacco cessation, and the risk of developing a second primary lung cancer.
  Arms: Lung Cancer Screening Education Group
Behavioral: Semi-Structured Interview — Participants will undergo an annual, in-person or virtual, semi-structured interviews to understand barriers and perception towards screening and cultural competencies to increase adherence to lung cancer screening. The interviews will last approximately 30 minutes at each visit.
  Arms: Lung Cancer Screening Education Group
Behavioral: Standard of Care Lung Cancer Screening Program — Participants will receive standard of care referral to the University of Miami's Lung Cancer Screening Program. The standard education includes a one-time, in-person or virtual 60-minute visit with the Advanced Practice Registered Nurse (APRN) to review educational material about lung cancer screening and tobacco cessation guidelines, and to discuss the risks versus benefits of undergoing screening.

SUMMARY:
The purpose of this study is to assess the awareness of eligibility of lung cancer screening in Hispanic/LatinX Head and Neck Cancer (HNC) survivors using a survey questionnaire; and to understand the barriers to screening using qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand, and sign informed consent form.
* Age ≥ 18 years.
* Participants must self-identify as Hispanic/LatinX.
* Individuals must be head and neck cancer survivors (treated locally with surgery, radiation alone, or definitive chemoradiation ≥ 5 years earlier and have no signs/symptoms to suggest recurrence of disease).
* Subjects that meet lung cancer (LC) screening eligibility according to United States Preventive Services Task Force (USPSTF21) and/or National Comprehensive Cancer Network (NCCN). For patients with a history of head and neck cancers, the NCCN recommends annual screening with low dose computerized tomography (LDCT) in those who have had a history of 20 pack years of smoking or more. USPSTF21 LC screening eligibility includes adults ages 50-80 that are current smoker or former smokers that quit within 15 years and have a 20 pack-year history or more of smoking.

Exclusion Criteria:

* Individuals with pre-established diagnosis of lung cancer.
* Participants with current diagnosis of any active malignancy.
* Subjects that had undergone lung imaging within previous 3 years.
* Pregnant or nursing mothers.
* Individuals that received head and neck related treatment less than 5 years before screening.
* Individuals with < 20 pack year history of smoking.
* Subjects with previous history of distant metastatic head and neck cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants' awareness of the risk of second primary lung cancer as measured by the University of Miami lung cancer screening program survey questionnaire. | Up to 2 Years
  The proportion of participants' awareness of the risk of second primary lung cancer will be assessed via the University of Miami lung cancer screening program survey questionnaire. Awareness of the risk of second primary lung cancer will be reported as the proportion of participants that indicated 'Yes' and 'No' on the survey questionnaire.
Proportion of participants' awareness of lung cancer screening recommendations as measured by the University of Miami lung cancer screening program survey questionnaire. | Up to 2 Years
  The proportion of participants' awareness of lung cancer screening recommendations will be assessed via the University of Miami lung cancer screening program survey questionnaire. Awareness of the lung cancer screening recommendations will be reported as the proportion of participants that indicated 'Yes' and 'No' on the survey questionnaire.
Proportion of participants' perception of the risk of second primary lung cancer as measured by the University of Miami lung cancer screening program survey questionnaire. | Up to 2 Years
  The proportion of participants' perception of the risk of second primary lung cancer will be assessed via the University of Miami lung cancer screening program survey questionnaire. Perception of the risk of second primary lung cancer will be reported as the proportion of participants that indicated 'Yes' and 'No' on the survey questionnaire.
Proportion of participants' perception of lung cancer screening recommendations as measured by the University of Miami lung cancer screening program survey questionnaire. | Up to 2 Years
  The proportion of participants' perception of lung cancer screening recommendations will be assessed via the University of Miami lung cancer screening program survey questionnaire. Perception of the lung cancer screening recommendations will be reported as the proportion of participants that indicated 'Yes' and 'No' on the survey questionnaire.

SECONDARY OUTCOMES:
Change in proportion of participants that undergo early detection lung cancer screening | Baseline, 1 Year
  The change in the proportion of participants that undergo early detection lung cancer screening will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Coral Olazagasti, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No